CLINICAL TRIAL: NCT04970186
Title: Assessment of Anatomical Variations of Greater Palatine Foramen in a Sample of Egyptian Population Using CBCT: A Hospital-based Cross-Sectional Study
Brief Title: Assessment of Anatomical Variations of Greater Palatine Foramen in a Sample of Egyptian Population (CBCT)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farid Medhat, principal investigator, Cairo University
Other Study IDs: ORAD 7-1-1
Record Dates: First submitted 2021-07-11; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Greater Palatine Foramen
Keywords: Greater palatine foramen; GPF; CBCT; Cone beam computed tomography; Hard palate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study to assess the anatomical variations of greater palatine foramen in a sample of Egyptian population using cone beam computed tomography through retrospective data analysis

DETAILED DESCRIPTION:
A) Setting and location:

1. The CBCT Scans of this study will be obtained from the data base available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University, Cairo, Egypt.
2. Being a retrospective study, CBCT scans of Egyptian patients who have already been subjected to CBCT examination as part of their dental diagnosis and/or treatment planning will be included according to the proposed eligibility criteria.

B)Participants:

Based on sample size calculation, a sample of 173 hemi-palate belonging to Egyptian individuals will be examined.

C) Variables:

* Details about variable

  1. Diameter of GPF.
  2. Location of GPF in relation to maxillary molars.
  3. The distance between the GPF and the midline maxillary suture (MMS).
  4. The distance between the GPF and the posterior border of the hard palate (PB).
  5. Number of foramina.
  6. Type of the hard palate and relation to GPF location:
* Palatal index
* Palatal height index

D)Data sources/ Measurements:

* Retrospective Data collection will be performed after the CBCT scans are pooled from the computer database.
* All the CBCT examinations will be scanned using CBCT machine (Planmeca promax 3D Mid).
* CBCT scans using different fields of view, with 0.4mm voxel size.
* The following parameters will be measured on these images in sagittal, coronal and axial planes:

  1. Diameter of GPF.
  2. Location of GPF in relation to maxillary molars as described by Ajmani (1994). Between the upper first and second molar - A In the midline of the upper second molar - B Between the upper second and third molar - C In the midline of the upper third molar - D Distal to the upper third molar - E
  3. The distance between the GPF and the midline maxillary suture
  4. The distance between the GPF and the posterior border of the hard palate (PB).
  5. Number of GPF.
  6. Type of the hard palate and relation to GPF location:
* Palatal index
* Palatal height index
* CBCT scans will be interpreted by two oral radiologists independently; blinded from demographic data of the patients and from the results of each other.
* One of them will evaluate the images twice with a period of two weeks between the two reading sessions.
* Then inter-observational and intra-observational reliability between the observers will be evaluated.

E) Addressing potential sources of bias:

No source of bias. CBCT scans will be coded and interpreted by two oral and maxillofacial radiologists independently blinded from demographic data of the patients and from the results of each other.

F) Study Size:

The aim of the study is to assess the diameter and location of the greater palatine foramen in a sample of Egyptian population. Based upon the results of Ikuta, Carla Renata Sanomiya, et al 2013, the diameter of greater palatine foramen= 3.1 mm (±0.47). Acceptable margin of error=7%, a total sample size of 173 hemi-palate will be sufficient. Sample size calculation was performed using Benchmark Six Sigma.

G) Sampling strategy: The sample will be collected by convenience sampling.

H) Quantitative variables:

Subgrouping will be created to assess the variables regarding the gender and side.

1. Diameter of GPF.
2. Location of GPF in relation to maxillary molars.
3. The distance between the GPF and the midline maxillary suture (MMS).
4. The distance between the GPF and the posterior border of the hard palate (PB).
5. Number of foramina.
6. Type of the hard palate and relation to GPF location:

   * Palatal index
   * Palatal height index

I) Statistical methods:

Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans of Adult Egyptian population older than 18 years.
* CBCT scans showing the floor of the maxillary sinus.
* No artifacts in the maxillary region, which will affect the quality of the image

Exclusion Criteria:

* CBCT sans of completely edentulous maxilla.
* Patients with trauma, craniofacial surgery, orthognathic surgery and malignancies involving the maxillofacial region.
* Patients with cleft palate and other craniofacial anomalies.
* Dental implants in the alveolar region of premolars and molars due to artifacts.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Egyptian Population
Sampling Method: Non-Probability Sample
Enrollment: 173 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Diameter of GPF | one year
  Measuring device is CBCT Software on Planmeca Promax 3D Mid, Measuring unit is mm

SECONDARY OUTCOMES:
Location of GPF in relation to maxillary molars. | one year
  Measuring device is CBCT Software on Planmeca Promax 3D Mid, Measuring unit is percentage %

OTHER OUTCOMES:
The distance between the GPF and the midline maxillary suture (MMS). | one year
  Measuring device is CBCT Software on Planmeca Promax 3D Mid, Measuring unit is mm
The distance between the GPF and the posterior border of the hard palate (PB). | one year
  Measuring device is CBCT Software on Planmeca Promax 3D Mid, Measuring unit is mm
Number of foramina. | one year
  Measuring device is CBCT Software on Planmeca Promax 3D Mid, Measuring unit is score
Type of the hard palate and relation to GPF location: • Palatal index • Palatal height index | one year
  Measuring device is CBCT Software on Planmeca Promax 3D Mid, Measuring unit is percentage %